CLINICAL TRIAL: NCT00639171
Title: Clinical Implementation and Evaluation of MR Spectroscopy for Breast Cancer Detection
Brief Title: Evaluate the Use of the Magnetic Resonance Spectroscopy in Determining if the Breast Tumor is Benign or Malignant
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Andrzej Krol, PhD, State University of New York - Upstate Medical University
Other Study IDs: SUNYUMU 4909
Record Dates: First submitted 2008-03-12; First posted 2008-03-20 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Tumors
Keywords: breast; diagnostic radiology; suspicious breast tumors; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Subjects with suspicious breast lesions that warrant further evaluation will be followed to determination and confirmation of diagnosis.
- 2: Normal subjects used to evaluate software and to develop and optimize MR sequences will be examined.

SUMMARY:
Magnetic Resonance Spectroscopy (MRS) is a novel imaging technique for noninvasive probing of biochemical properties of tissue. While MRS does not generate images of tumor per se it allows biochemical spectroscopic data to be obtained in vivo from user defined region-of-interest. In this manner, biochemical information elucidated by MRS can be interpreted in relation to detailed anatomy and images of metabolite distribution can be created. The aim of MRS is to identify presence and concentration of metabolites characteristic for normal and abnormal (tumor) cellular activities hence allow differential normal tissue from pathological tissue, as well as allow differentiating malignant from benign tumors.

DETAILED DESCRIPTION:
Recent in vivo studies have reported successful use of 1H and 31P MRS in differentiating between benign and malignant tumors in breast tissue. These studies demonstrated an increase in the choline metabolite peak that reflects an increase in choline-containing metabolites in 70-80% of breast carcinomas, as compared to 14-18% of benign breast tumors.The objectives would be to determine sensitivity/specificity of MRS in the context of breast CA, We will use normal volunteers to test software and to develop and optimize MR scan sequences prior to or during the testing of target subjects with suspicious breast lesion.

ELIGIBILITY:
Inclusion Criteria:

* subjects should have well defined suspicious breast lesion and that will be biopsied
* subjects are to include; varied volunteers with different breast tissue with characteristics such as dense breasts, fibrocystic breasts, "small" breasted and "large" breasted women.

Exclusion Criteria:

* Women of childbearing potential who are not practicing a medically accepted method of birth control should not participate
* Subjects that are pregnant, breast-feeding, should not be able to participate
* Subjects having any of the following metallic devices, will be ineligible to participate in the study: pacemaker, prosthesis, artificial heart valve, coronary artery stents, TENS (Transcutaneous electric nerve stimulator) or other neurological stimulation units and surgical clips.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from two ongoing clinical studies of the breast at SUNY Upstate Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Krol, PhD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No